CLINICAL TRIAL: NCT04881370
Title: Quality of Life for Patients With Chronic Paediatric Onset Inflammatory Bowel Disease (IBD)
Acronym: QALY-ECOPED
Status: Terminated | Type: Observational
Why Stopped: insufficiency inclusion during the inclusion periode
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020_70; 2020-A00464-35 (Other: ID-RCB number, ANSM); PRME-15-0464 (Other: DGOS number, PRME number)
Record Dates: First submitted 2021-05-03; First posted 2021-05-11 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of the present study is to describe the quality of life of patients under 25 years of age with pediatric-onset IBD. The quality of life will be described according to the age and the activity of the disease in order to make it possible to associate with the different states of health a measure of quality of life (utility score) from utility values established in the French context. These data are essential for the realization of medico-economic models.

DETAILED DESCRIPTION:
The continuous increase in incidence of chronic inflammatory bowel disease (IBD) will increase their burden on health care costs in the future. Pediatric IBD is frequently associated with an aggressive phenotype causing specific complications (undernutrition, pubertal delay or height-weight loss) and has a long-term impact on quality of life.

Therapeutic evolutions were marked in the 1990s by the arrival of immunosuppressants and then in the 2000s of biotherapies (anti-TNF).To limit the accumulation of tissue damage and to benefit from the maximum effectiveness of anti -TNF, clinicians are tempted to offer early treatment of CD with anti-TNF.

An ongoing study using data from the EPIMAD registry aims to study the impact of therapies on the disease course of patients with IBD in their childhood (Inspired study). This study also contains a medico-economic component, the objective of which is to evaluate the cost-effectiveness of the different management strategies for pediatric onset IBD. As part of this economic study, quality of life data will be needed. Indeed, there are very few data on quality of life in children / adolescents with IBD in the literature. These data must be collected from patients, unlike the other data used (retrospective data, in medical records).

The main objective of the present study is to describe the quality of life of patients under 25 years of age with pediatric-onset IBD. The quality of life will be described according to the age and the activity of the disease in order to make it possible to associate with the different states of health a measure of quality of life (utility score) from utility values established in the French context. These data are essential for the realization of medico-economic models.

This study will supplement data currently being collected from patients over 25 years of age, quality of life being the subject of a secondary objective of a study on the professional integration of patients with IBD (PROMICI study , ID-RCB: 2017-A03397-46).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, between 12 and 24 years old included at the time of the study
* Subject listed in the EPIMAD registry suffering from certain or probable Crohn's disease, or certain or probable ulcerative colitis, or certain or probable ulcerative proctitis
* Disease diagnosed before the age of 17 (pediatric onset disease)
* Patient residing in the area of the EPIMAD register at the time of diagnosis: Nord, Pas-de-Calais, Somme or Seine-Maritime
* Patient not opposing the research
* Patient not having objected to the use of these data for ancillary studies when registering in the EPIMAD register

Exclusion Criteria:

* No exclusion criteria

Ages: 12 Years to 24 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients with pediatric-onset IBD (diagnosed before the age of 17) and aged over 12 and under 25 at the time of the study.
Sampling Method: Non-Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
Quality of life according to age and disease activity | through study completion, an average of 1 year
  Quality of life is measured by EQ5D-5L questionnaire and transformed into utility according to French reference values

SECONDARY OUTCOMES:
Correlation between EQ5D-5L and SIBDQ questionnaire in adults | through study completion, an average of 1 year
  EQ5D-5L is a generic measure of quality of life and SIBDQ a disease-specific questionnaire of quality of life
Correlation between EQ5D-5L and IMPACT III questionnaire in adolescents | through study completion, an average of 1 year
  EQ5D-5L is a generic measure of quality of life and IMPACT III a disease-specific questionnaire of quality of life
Quality of life according to previous surgery occurence | through study completion, an average of 1 year
  Quality of life is measured by EQ5D-5L
Correlation between quality of life and perceived health | through study completion, an average of 1 year
  Quality of life measured by EQ5D-5L and perceived health by Visual Analogue Scale
Quality of life according to profession and academic degree (adults only) | through study completion, an average of 1 year
  Quality of life as measured by EQ5D-5L
Quality of life according to profession and academic degree (adults only) | through study completion, an average of 1 year
  Quality of life as measured by SIBDQ

CONTACTS AND LOCATIONS:
Overall Officials: Dominique TURCK, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Jeanne de Flandre Chu Lille, Lille, France